CLINICAL TRIAL: NCT02074293
Title: ASIS for Botox in Cervical Dystonia
Acronym: ASISinCD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: li nguyen (Industry)
Responsible Party: Sponsor-Investigator, li nguyen, MD/CEO/PI, ASIS Corporation
Organization: ASIS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCTNS089268; R44NS089268 (Other Grant/Funding Number: NATIONAL INSTITUTE OF NEUROLOGICAL DISORDERS AND STROKE)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Dystonia Adults ,; Abnormal Head Position and Neck Pain for These 7 Muscle Groups: Splenius,Scalene,Sterno-cleido-mastoid,Levator Scapulae,Semispinalis,Trapezius,and Longissimus.
Keywords: Subdermal bloodless space; Subdermal injection; injectable EMG needle; electrical stimulation; MRI with Gadolinium; Cervical Dystonia; intramuscular injection; cervical dystonia,
MeSH Terms: conditions — Torticollis | interventions — Gadolinium; Gadolinium DTPA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (22):
- Splenius (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Scalene (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Sterno-cleido-mastoid (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Levator Scapulae (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Semispinalis (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Trapezius (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Longissimus (Experimental): Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9ccNS intramuscularly for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- Change from Baseline in Pain Frequency (Experimental): Change from Baseline in Pain Frequency as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30.
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in Pain Intensity (Experimental): Change from Baseline in Pain Intensity as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. The severity on scales of 0(no pain) to 4(constant or extremely severe intensity).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Change from Baseline in CDSS (Experimental): Change from Baseline in CDSS as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. The CDSS or Cervical Dystonia Severity Scale quantifies the severity of abnormal head positioning and was newly devised for this study. CDSS allots 1 point for each 5 degrees (or part thereof) of head deviation in each of the three planes of head movement (range of scores up to theoretical maximum of 54).
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Percent of Patients with Improved PGAS (Experimental): Percent of Patients with Improved PGAS as Efficacy of Botox intramuscularly at Week 6, Efficacy of Botox intramuscularly at Week 12, Efficacy of Botox intramuscularly at Week 18, Efficacy of Botox intramuscularly at Week 24, and Efficacy of Botox intramuscularly at Week 30 vs.Efficacy of Botox subdermally at Week 6, Efficacy of Botox subdermally at Week 12, Efficacy of Botox subdermally at Week 18, Efficacy of Botox subdermally at Week 24, and Efficacy of Botox subdermally at Week 30. The Physician Global Assessment Scale or PGAS is a 9 category scale scoring the physician's evaluation of the patients' status compared to baseline, ranging from -4 to +4 (very marked worsening to complete improvement), with 0 indicating no change from baseline and +1 slight improvement.
  Interventions: Drug: Efficacy of Botox intramuscularly at Week 6; Drug: Efficacy of Botox intramuscularly at Week 12; Drug: Efficacy of Botox intramuscularly at Week 18; Drug: Efficacy of Botox intramuscularly at Week 24; Drug: Efficacy of Botox intramuscularly at Week 30; Drug: Efficacy of Botox subdermally at Week 6; Drug: Efficacy of Botox subdermally at Week 12; Drug: Efficacy of Botox subdermally at Week 18; Drug: Efficacy of Botox subdermally at Week 24; Drug: Efficacy of Botox subdermally at Week 30
- Adverse Reactions with Facial paresis (Experimental): Facial paresis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Eyelid ptosis (Experimental): Eyelid ptosis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Bronchitis (Experimental): Bronchitis as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Neck pain (Experimental): Neck pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle stiffness (Experimental): Musculoskeletal stiffness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscular weakness (Experimental): Muscular weakness as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Myalgia (Experimental): Myalgia as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle pain (Experimental): Musculoskeletal pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Muscle spasms (Experimental): Muscle spasms as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions Injection site pain (Experimental): Injection site pain as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally
- Adverse Reactions with Hypertension (Experimental): Hypertension as Adverse Reactions of Botox intramuscularly vs.Adverse Reactions of Botox subdermally at Week 30.
  Interventions: Drug: Adverse Reactions of Botox intramuscularly; Drug: Adverse Reactions of Botox subdermally

INTERVENTIONS:
Drug: Gadolinium — Gadolinium .1cc/ diluted with .9ccNS intramuscularly with ASIS Device for 30 patients. Total cumulative Persistent % of Gadolinium intramuscularly on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Levator Scapulae; Longissimus; Scalene; Semispinalis; Splenius; Sterno-cleido-mastoid; Trapezius
Drug: Gadolinium — Gadolinium .1cc/ diluted with .9ccNS subdermally with ASIS Device for 30 patients. Total cumulative Persistent % of Gadolinium subdermally on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Levator Scapulae; Longissimus; Scalene; Semispinalis; Splenius; Sterno-cleido-mastoid; Trapezius
Drug: Gadolinium — Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium intramuscularly on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: Levator Scapulae; Longissimus; Scalene; Semispinalis; Splenius; Sterno-cleido-mastoid; Trapezius
Drug: Efficacy of Botox intramuscularly at Week 6 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 6, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox intramuscularly at Week 12 — Efficacy of Botox intramuscularly at Week 12, in terms of Percent of Patients with Improved PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, Change from Baseline in Pain Intensity, Change from Baseline in CDSS (Cervical Dystonia Severity Scale).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox intramuscularly at Week 18 — Efficacy of Botox intramuscularly at Week 18, in terms of Percent of Patients with Improved PGAS, or improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, Change from Baseline in Pain Intensity, Change from Baseline in CDSS (Cervical Dystonia Severity Scale).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox intramuscularly at Week 24 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 24, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox intramuscularly at Week 30 — Efficacy of Botox (onabotulinumtoxinA) intramuscularly at Week 30, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox subdermally at Week 6 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 6, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox subdermally at Week 12 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 12, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox subdermally at Week 18 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 18, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox subdermally at Week 24 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 24, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Efficacy of Botox subdermally at Week 30 — Efficacy of Botox (onabotulinumtoxinA) subdermally at Week 30, in terms of improvement on the Physician Global Assessment Scale, and Change from Baseline in Pain Frequency, and Pain Intensity, as well as Cervical Dystonia Severity Scale (CDSS).
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Change from Baseline in CDSS; Change from Baseline in Pain Frequency; Change from Baseline in Pain Intensity; Percent of Patients with Improved PGAS
Drug: Adverse Reactions of Botox intramuscularly — Adverse Reactions of Botox (onabotulinumtoxinA) intramuscularly at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain
Drug: Adverse Reactions of Botox subdermally — Adverse Reactions of Botox (onabotulinumtoxinA) subdermally at Week 30, in number of Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.
  Other Names: Botox (onabotulinumtoxinA)
  Arms: Adverse Reactions Injection site pain; Adverse Reactions with Bronchitis; Adverse Reactions with Eyelid ptosis; Adverse Reactions with Facial paresis; Adverse Reactions with Hypertension; Adverse Reactions with Muscle pain; Adverse Reactions with Muscle spasms; Adverse Reactions with Muscle stiffness; Adverse Reactions with Muscular weakness; Adverse Reactions with Myalgia; Adverse Reactions with Neck pain

SUMMARY:
Botox acts on nerve endings, yet there are no nerve endings inside the muscle, where they are typically injected. All nerves terminate on the fascia, where ASIS device can precisely deliver Botox by creating that subdermal bloodless space, between the skin and muscle. Thus enhancing and prolonging Botox's efficacy, at the same time prevent it's unnecessary adverse reactions and distant spread, especially since Botox has no reason to travel to the rest of the body any way.

DETAILED DESCRIPTION:
Aim 1 over 6 months will demonstrate ASIS device's consistent performance on 60 adult subjects with Cervical Dystonia. Gadolinium will be injected with ASIS subdermally (30) or conventional intramuscularly (30) for these 7 muscle groups: Splenius, Scalene, Sterno-cleido-mastoid, Levator scapulae, Semispinalis, Trapezius, and Longissimus. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. Since there isn't a way to measure level of Gadolinium within it, or any other (e.g. Botox) for that matter, at least the Prolongation of Gadolinium may be approximated by the greater or longer Persistent % on MRI. However, this approximation can only work if the variables are minimized to the same population with Cervical Dystonia, and these particular 7 muscle groups. Case in point, patients with Cervical Dystonia presumably have hyperactive Splenius, Scalene, Sterno-cleido-mastoid, Levator scapulae, Semispinalis, Trapezius, and Longissimus muscles, so expectantly will have shortened Gadolinium intramuscularly Persistent %, and somewhat reduced Gadolinium subdermally Persistent % as well due to agitation, thus these Persistent % values in Cervical Dystonia patients will not be like those of normal patients, or even the same between these 7 different muscle groups. Therefore, the Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, will be specific and valuable indicators to help us modify Botox dosage and duration to inject into "unknown" subdermal bloodless space for Aim 2.

Aim 2 over 12 months, using Botox, instead of Gadolinium, will demonstrate the advantages of ASIS device subdermally over intramuscularly, for the same 60 adult subjects with Cervical Dystonia, on these particular 7 muscle groups: Splenius, Scalene, Sterno-cleido-mastoid, Levator scapulae, Semispinalis, Trapezius, and Longissimus. Hypothetically speaking, if that subdermal bloodless space in patients with e.g., Cervical Dystonia somehow failed to show prolongation of half-life for Gadolinium in Aim 1, we can still proceed with primary interest being therapeutic comparison for Botox in Aim 2, in terms of improvement on the Physician Global Assessment Scale at 6, 12, 18, 24, and 30 weeks, and reduction in Cervical Dystonia Severity Scale (CDSS) as well as adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

•Adults with cervical dystonia, or abnormal head position and neck pain for these 7 muscle groups: Splenius, Scalene, Sterno-cleido-mastoid, Levator scapulae, Semispinalis, Trapezius, and Longissimus.

Exclusion Criteria:

* Known Hypersensitivity to Botulinum Toxin or to any of the components in the formulation.
* Infection at the Injection Site(s).
* Has any medical condition that may increase their risk with exposure to Botox including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.
* Has profound atrophy or weakness of muscles in the target areas of injection.
* Had previously received surgical or other denervation treatment for their symptoms or had a known history of neuromuscular disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative Prolongation Ability Score for Gadolinium subdermally injected. | 6 months
  Gadolinium will be injected with ASIS subdermally (30) or conventional intramuscularly (30) in Cervical Dystonia adult patients for these 7 muscle groups: Splenius, Scalene, Sterno-cleido-mastoid, Levator scapulae, Semispinalis, Trapezius, and Longissimus. An MRI will be taken promptly after Gadolinium injection, as starting reference, to which subsequent MRI taken at 6 hrs, 12 hrs, and 24 hrs later will be compared for Persistent %. This approximation can only work if the variables are minimized to the same population with Cervical Dystonia, and these particular 7 muscle groups. The Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % intramuscularly, in Cervical Dystonia patients will not be like those of normal patients, or even the same between these 7 different muscle groups, but valuable indicators to help us modify Botox dosage and duration to inject into "unknown" subdermal bloodless space for Aim 2.

SECONDARY OUTCOMES:
Efficacy of Botox intramuscularly vs. subdermally in Cervical Dystonia. | 12 months
  Efficacy of Botox intramuscularly vs. subdermally with ASIS Device at Week 6,12,18, 24, and 30; in terms of improvement on the Physician Global Assessment Scale (-4=very marked worsening to +4=very marked improvement). Also in terms of improvement, or Median Change from Baseline in Pain Frequency, Pain Intensity (0(no pain) to 4(constant or extremely severe intensity)), and Cervical Dystonia Severity Scale (CDSS). CDSS allots 1 point for each 5 degrees (or part thereof) of head deviation in each of the three planes of head movement (range of scores up to theoretical maximum of 54).

OTHER OUTCOMES:
Adverse Reactions of Botox intramuscularly vs. subdermally in Cervical Dystonia. | 12 months
  Adverse Reactions of Botox intramuscularly vs. subdermally:
  Headache Migraine, Facial paresis, Eyelid ptosis, Bronchitis, Neck pain Musculoskeletal stiffness, Muscular weakness Myalgia, Musculoskeletal pain, Muscle spasms, Injection site pain, and Hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- Automatic Subdermal Injector System, Inc, Westminster, California, United States

REFERENCES:
- [Background] Lorenc ZP, Kenkel JM, Fagien S, Hirmand H, Nestor MS, Sclafani AP, Sykes JM, Waldorf HA. A review of onabotulinumtoxinA (Botox). Aesthet Surg J. 2013 Mar;33(1 Suppl):9S-12S. doi: 10.1177/1090820X12474629. PMID 23515199
- [Background] Knopp MV, Balzer T, Esser M, Kashanian FK, Paul P, Niendorf HP. Assessment of utilization and pharmacovigilance based on spontaneous adverse event reporting of gadopentetate dimeglumine as a magnetic resonance contrast agent after 45 million administrations and 15 years of clinical use. Invest Radiol. 2006 Jun;41(6):491-9. doi: 10.1097/01.rli.0000209657.16115.42. PMID 16763467
- [Background] Velickovic M, Benabou R, Brin MF. Cervical dystonia pathophysiology and treatment options. Drugs. 2001;61(13):1921-43. doi: 10.2165/00003495-200161130-00004. PMID 11708764
- [Background] Claypool DW, Duane DD, Ilstrup DM, Melton LJ 3rd. Epidemiology and outcome of cervical dystonia (spasmodic torticollis) in Rochester, Minnesota. Mov Disord. 1995 Sep;10(5):608-14. doi: 10.1002/mds.870100513. PMID 8552113
- [Background] Tiderington E, Goodman EM, Rosen AR, Hapner ER, Johns MM 3rd, Evatt ML, Freeman A, Factor S, Jinnah HA. How long does it take to diagnose cervical dystonia? J Neurol Sci. 2013 Dec 15;335(1-2):72-4. doi: 10.1016/j.jns.2013.08.028. Epub 2013 Aug 30. PMID 24034410
- [Background] Albanese A, Sorbo FD, Comella C, Jinnah HA, Mink JW, Post B, Vidailhet M, Volkmann J, Warner TT, Leentjens AF, Martinez-Martin P, Stebbins GT, Goetz CG, Schrag A. Dystonia rating scales: critique and recommendations. Mov Disord. 2013 Jun 15;28(7):874-83. doi: 10.1002/mds.25579. PMID 23893443
- [Background] Evidente VG, Fernandez HH, LeDoux MS, Brashear A, Grafe S, Hanschmann A, Comella CL. A randomized, double-blind study of repeated incobotulinumtoxinA (Xeomin((R))) in cervical dystonia. J Neural Transm (Vienna). 2013 Dec;120(12):1699-707. doi: 10.1007/s00702-013-1048-3. Epub 2013 Jun 19. PMID 23779062
- [Background] Leplow B, Bottcher M, Schonfeld R. [Botulinum toxin therapy for spasmodic torticollis: medical and non-medical adjunct treatment]. Nervenarzt. 2013 Apr;84(4):493-7. doi: 10.1007/s00115-012-3708-1. German. PMID 23371379
- [Background] Vivancos-Matellano F, Ybot-Gorrin I, Diez-Tejedor E. A 17-year experience of abobotulinumtoxina in cervical dystonia. Int J Neurosci. 2012 Jul;122(7):354-7. doi: 10.3109/00207454.2012.665971. Epub 2012 Mar 20. PMID 22329596
- See also: Click here for more information about this study ASIS for Botox in Cervical Dystonia — http://www.asis-inc.com